CLINICAL TRIAL: NCT01416844
Title: Phase II Exploratory Study of Immune Responses in Patients With Metastatic Melanoma Treated With Mouse Monoclonal Anti-OX40
Brief Title: Study of Immune Responses in Patients With Metastatic Melanoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Change in the development plan for the anti-OX40 antibody.
Sponsor: Providence Health & Services (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PH&S IRB 10-090
Record Dates: First submitted 2011-08-12; First posted 2011-08-15 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-03

CONDITIONS: Metastatic Melanoma
Keywords: Metastatic melanoma; anti-OX40; Immunostimulatory
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: anti-OX40 — Patients with metastatic melanoma will be given 0.4 mg/kg anti-OX40 on days 1, 3 and 5 of a single treatment cycle.

SUMMARY:
In this study, anti-OX40 will be given to patients with melanoma to find out how the immune system responds to treatment with anti-OX40. It is hoped that this treatment will cause an immune response against melanoma resulting in tumor regression, but this is not known at this time. Anti-OX40 is a large protein that can help immune cells that fight bacteria, viruses and cancer cells.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with measurable or evaluable unresectable, stage IV metastatic melanoma. Either histologic or cytologic diagnosis is acceptable.
2. Eastern Cooperative Oncology Group (ECOG) performance status 0, or 1 (Appendix A.)
3. Age 18 years or above.
4. Laboratory values (performed within 28 days prior to enrollment) as follows:

   * WBC ≥2000/microliter
   * Absolute lymphocyte count >300/mm3
   * Serum creatinine <1.5 X upper limit of laboratory normal
   * Hgb >8g/dl (patients may be transfused to reach this level)
   * Hct > 24%
   * Platelets >100,000 cells/mm3
   * Total bilirubin <1.5 X upper limit of laboratory normal, unless due to Gilbert's disease
   * AST (SGOT)/ALT (SGPT) <2.5 X upper limit of laboratory normal
   * Alkaline phosphatase <2.5 X upper limit of laboratory normal
   * HIV Negative
   * Hepatitis B surface antigen Negative
   * Hepatitis C antibody Negative
5. Women of childbearing potential must have a negative pregnancy test and must avoid becoming pregnant while on treatment. Men must avoid fathering a child while on treatment. This exclusion is required due to the unknown toxicities that anti-OX40 may have on the forming fetus, spermatogenesis or the nursing child. Also, because pregnancy may impair immune function it may limit the treatment efficacy.
6. Ability to give informed consent and comply with the protocol. Patients with a history of psychiatric illness must be judged able to understand fully the investigational nature of the study and the risks associated with the therapy.
7. No active bleeding.
8. No clinical coagulopathy (INR <1.5, PT <16 seconds, PTT < 38 seconds).
9. Anticipated lifespan greater than 12 weeks.
10. Failed at least one prior medical therapy for metastatic melanoma.

Exclusion Criteria:

1. Active infection.
2. History of or active autoimmune disease.
3. Prior mouse monoclonal antibody treatment.
4. Pregnant or lactating women, as treatment involves unforeseeable risks to the embryo or fetus.
5. Need for chronic maintenance oral steroids.
6. Active brain metastatic disease. Treated brain metastases with surgery, gamma-knife radiosurgery and/or whole brain radiation and stable for at least 4 weeks and off steroids are eligible.
7. Any medical or psychiatric condition that in the opinion of the PI would preclude compliance with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Increased number of tumor antigen specific circulating T Cells | Screening (baseline) and Day 15
  T Cells will be harvested by apheresis at baseline and Day 15 following anti-OX40 administration.

CONTACTS AND LOCATIONS:
Overall Officials: Brendan D Curti, MD, Principal Investigator — Providence Health & Services
Locations (1):
- Providence Portland Medical Center, Portland, Oregon, United States